CLINICAL TRIAL: NCT06808932
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose (SAD) Study With Food-Effect Cohort to Assess the Safety, Tolerability, and Pharmacokinetics of Oral (R) VK4-116 in Healthy Volunteers
Brief Title: VK4-116 Phase I Study With Food-Effect
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-VK4-116-Ph1a-001
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Opioid Dependence; Opioid Use Disorder (OUD)
Keywords: addiction; dopamine; dopamine receptor
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive | interventions — VK4-116

STUDY DESIGN:
Intervention Model Description: This is first-in-human (FIH), randomized, double-blind, placebo-controlled, single ascending dose (SAD), phase I study in healthy participants. Five single ascending dose levels under fasting conditions are proposed. This study will also provide a preliminary assessment of the potential effect of food on the dose corresponding to approximately 40% of the maximum safe and well-tolerated dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- 50 mg dose (Experimental): oral administration in fasted state
  Interventions: Drug: VK4-116
- 100 mg dose (Experimental): oral administration in fasted state
  Interventions: Drug: VK4-116
- 200 mg dose (Experimental): oral administration in fasted state
  Interventions: Drug: VK4-116
- 400 mg dose (Experimental): oral administration in fasted state
  Interventions: Drug: VK4-116
- 500 mg dose (Experimental): oral administration in fasted state
  Interventions: Drug: VK4-116
- 200 mg dose in fed state (Experimental): oral administration in fed state
  Interventions: Drug: VK4-116
- placebo (Placebo Comparator): oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VK4-116 — D3R antagonist
  Arms: 100 mg dose; 200 mg dose; 200 mg dose in fed state; 400 mg dose; 50 mg dose; 500 mg dose
Drug: Placebo — Each of the four dose groups of n=8 participants will be assigned to active drug or placebo in the ration 6:2.
  Arms: placebo

SUMMARY:
This first-in-human, randomized, double-blind, placebo-controlled, single ascending dose (SAD), phase I study is designed to assess the safety, tolerability and pharmacokinetics of VK4-116 in healthy volunteers in fasted and fed state.

DETAILED DESCRIPTION:
Approximately 48 healthy volunteers will be enrolled and randomized to receive either VK4-116 or a placebo within one of five ascending dose cohorts. Each cohort will consist of eight participants, with a 6:2 ratio of active drug to placebo assignment. Dose escalation decisions will be made following a review of blinded safety, tolerability, and pharmacokinetic (PK) data from the preceding cohort.

The proposed dose levels under fasting conditions are 50 mg, 100 mg, 200 mg, 400 mg, and 500 mg. Additional cohort will receive a 200 mg dose in a fed state, approximately 30 minutes after a high-fat, high-calorie breakfast. Dose adjustments may be made based on the safety, tolerability, and PK data observed in earlier cohorts.

Participants will be admitted to the research clinic one day prior to receiving their assigned treatment. Following the administration of VK4-116 or placebo, participants will be continuously monitored for adverse events, and PK blood samples will be collected at predetermined intervals. Participants will remain in the clinic for 4 days, until the 72-hour PK blood sample has been collected. Participants in the food-effect cohort will stay in the clinic for 8 days (for fasted stat followed by fed state assessments). A follow-up visit will be scheduled three days after discharge from the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy male or female volunteer between 18 and 60 years of age, inclusive, at the time of consent.

   • The masculine / feminine gender is used without any discrimination and with the aim to lighten the text.
2. Have a body mass index (BMI) within a range of 17.0 to 36.0 kg/m2 and a minimum weight of at least 50.0 kg at screening.
3. Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures.
4. Have no clinically significant concurrent medical conditions determined by medical history, physical examination, clinical laboratory examination, vital signs, and 12-lead ECG.
5. A female study participant must meet one of the following criteria:

   * If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first administration of the study medication, during the study, and for at least 30 days after the last dose of the study medication. An acceptable method of contraception includes one of the following:

     i. abstinence from heterosexual intercourse, ii. hormonal contraceptives (e.g., injectable/implant/insertable hormonal birth control products, transdermal patch), iii. intrauterine device (with or without hormones). OR agrees to use a double barrier method (e.g., condom and spermicide) during the study and for at least 30 days after the last dose of the study medication.
   * If a female of non-childbearing potential - should be surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses), as confirmed by follicle stimulating hormone (FSH) levels (≥40 mIU/mL).

   A male study participant that engages in sexual activity must agree to use a double barrier method (e.g., condom and spermicide) and agree to not donate sperm during the study and for at least 90 days after the last dose of the study medication.
6. Be able and willing to comply with protocol requirements and the rules and regulations of the study site, and be likely to complete all the study treatments.

Exclusion Criteria:

1. Have any clinically significant finding within one year of Screening on medical history, physical examination, complete neurological examination, clinical laboratory test, vital signs or ECGs that contraindicate participation in the study. This includes, but is not limited to, history of or current cardiac, hepatic, renal, neurologic, gastrointestinal (GI), pulmonary, endocrinologic, hematologic, or immunologic disease or history of malignancy.
2. Use nicotine products via smoking/vaping in past 6 months.
3. Have a sitting systolic blood pressure (BP) >140 mmHg, diastolic BP >90 mmHg and heart rate (HR) <45 or >100 beats per minute (BPM) at screening and clinic intake.
4. History of unstable angina; a history of myocardial infarction; or a history of a clinically significant cardiac arrhythmia,
5. Has a QT interval corrected for heart rate using Fredericia formula >450 milliseconds in males or >470 milliseconds in females, or evidence of left bundle branch blocks (Note: right bundle branch block is acceptable), second or third degree AV block, or evidence of left ventricular hypertrophy on ECG
6. Have a history of liver disease or current elevation of aspartate aminotransferase (AST), alanine aminotransferase (ALT), 2 × the upper limit of normal (ULN).
7. Have a history of renal disease or current renal function test values as follows:

   * blood urea nitrogen (BUN) >2 × ULN,
   * creatinine (Cr) >1.5 mg/dL.
8. Have donated blood (excluding plasma donation) of approximately 500 mL within 56 days prior to screening.
9. Have donated plasma within 7 days prior to screening.
10. Have hemoglobin value of <13 g/dL for men and <12 g/dL for women.
11. Have undergone treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to screening.
12. Have taken prescribed medications within 14 days of Day -1 or over-the-counter medications, dietary supplements, herbal products, or vitamins within 7 days or 5 half-lives (if known), whichever is longer, of Day -1.
13. Have a positive urine drug test for alcohol, opioids (e.g., codeine, heroin, fentanyl, morphine, oxycodone, etc.), cocaine, amphetamine, methamphetamine, 3,4-methylenedioxymethamphetamine (MDMA), benzodiazepines, tetrahydrocannabinol (THC), barbiturates, propoxyphene, or phencyclidine/phenylcyclohexyl piperidine (PCP) at admission.
14. Have a history of suicide attempts or current or recent evidence of suicidal ideation in the past 12 months based on the Columbia-Suicide Severity Rating Scale (C-SSRS).
15. Have a positive serology for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV).
16. Have positive results for a coronavirus disease 2019 (COVID-19) test.
17. Have a history of anaphylaxis and known allergy to any drug formulation.
18. Have a history of consumption of any product containing grapefruit, pomelo, Seville oranges, or alcohol within 7 days before study drug dosing on Day 1.
19. Have consumed any product containing caffeine or xanthine within 24 hours before study drug dosing on Day 1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events in Healthy Adult Participants | 7 days for fasted condition, 11 days for fed condition
  The incidence of treatment-emergent adverse events will be measured using a combination of data collection methods, including tracking adverse events and assessing their onset or worsening relative to the initiation of treatment. The most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) preferred terms will be used to classify adverse events, including their relationship to the treatment and maximum severity. Events will be identified either through subject self-report or clinically significant abnormal findings on:
  (i) Physical examination (ii) Vital signs assessments (heart rate (BPM), blood pressure (mmHg), respiration rate (BPM), and temperature (F)) (iii) ECG assessment (QTcF) as determined by the Investigator/consulting board-certified cardiologist (iv) Clinical Laboratory Assessments

SECONDARY OUTCOMES:
Cmax | 72 hours
  maximum observed plasma concentration (ng/mL)
AUC | 72 hours
  area under the concentration-time curve (mg*h/L)
Tmax | 72 hours
  time of maximum observed plasma concentration (hours)
half life (t½) | 72 hours
  VK4-116 elimination half-life (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Marta De Santis, PhD, Study Director — National Institute on Drug Abuse, NIH
Locations (1):
- Altasciences Clinical Kansas, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided